CLINICAL TRIAL: NCT02145403
Title: Phase 1/2 Study of Carfilzomib for the Prevention of Relapse and Graft-versus-host Disease in Allogeneic Hematopoietic Cell Transplantation for High-risk Hematologic Malignancies
Brief Title: Phase 1/2 Study of Carfilzomib for the Prevention of Relapse and GVHD in Allo-HCT for Hematologic Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2014.010; HUM00084170 (Other: University of Michigan)
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Results first posted 2020-01-06 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Hematologic Malignancies; Relapse; Graft-Versus-Host Disease
Keywords: Allogeneic Transplantation; Carfilzomib; Relapse; Graft-Versus-Host Disease; Multiple Myeloma; Lymphoma; Leukemia
MeSH Terms: conditions — Hematologic Neoplasms; Recurrence; Graft vs Host Disease; Multiple Myeloma; Lymphoma; Leukemia | interventions — carfilzomib; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carfilzomib (Experimental): Carfilzomib will be administered IV over 30 minutes, starting at dose level 1 (20 mg/m2 IV) on Day +1, +2, +6 and +7.
  Interventions: Drug: Carfilzomib; Drug: Tacrolimus

INTERVENTIONS:
Drug: Carfilzomib — Carfilzomib will be administered starting at dose level 1 (20 mg/m2 IV) on day +1, +2, +6 and +7.
  Dose escalation will be performed on the day +6 and day +7 doses only in each dose level. Day +1 and day+2 doses will be fixed at 20 mg/m2 IV in all dose levels.
  Other Names: Kyprolis®
Drug: Tacrolimus — Tacrolimus will be administered at 0.03 mg/kg continuous infusion over 24 hours, starting on day -3 as standard graft-versus-host disease prophylaxis.

SUMMARY:
The investigators hypothesize that adding carfilzomib to standard conditioning regimen for allo-HCT for advanced or high-risk hematologic malignancies will decrease post-transplant relapse and treatment-related mortality by decreasing severe GVHD, leading to overall improvement in transplant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Lymphoid or Myeloid malignancy requiring allogeneic hematopoietic cell transplantation
* Pathology review by the study institution is required
* Prior high-dose chemotherapy and autologous HCT(s) is (are) allowed
* Disease status: Stable disease or better at the time of enrollment
* Age: >18 and <70 years old at the time of transplant (< 71 years at transplant admission)
* Life expectancy ≥ 6 months after transplant
* A 8/8 or 7/8 HLA-matched donor is available
* Karnofsky Performance Status >70% (A measure of quality of life that ranges from 0 to 100 where 100 equals perfect health and 0 is death.)
* Adequate cardiac [LVEF (Left Ventricular Ejection Fraction) >0.4], pulmonary [FEV1 (Forced Expiratory Volume in 1 Second), FVC (Forced Vital Capacity), corrected DLCO (Diffusing Capacity) ≥ 50% predicted], hepatic [DB (Direct Bilirubin) <1.5xULN, AST (Aspartate Aminotransferase) / ALT (Alanine transaminase) ≤3xULN] and renal function [GFR (Glomerular Filtration Rate) ≥ 60 mL/min/1.73 m2]

Exclusion Criteria:

* Progressive disease
* Active central nervous system involvement by malignancy
* Non compliance to medications or medical instructions
* Lack of appropriate caregivers
* Life expectancy <6 months
* Pregnant or lactating females
* Uncontrolled infection requiring active treatment (systemic antibiotics, anti-virals, or anti-fungals) within 14 days
* HIV-1/HIV-2 or HTLV-1/HTLV-2 seropositivity
* Active hepatitis A, B or C infection
* Unstable angina or myocardial infarction within 6 months prior to randomization, NYHA Class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, uncontrolled or persistent atrial fibrillation/flutter, history of ventricular fibrillation, ventricular tachycardia/torsade de pointes, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker
* History of pulmonary hypertension
* Uncontrolled hypertension or uncontrolled diabetes mellitus
* Non-hematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen (PSA) levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas
* Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib)
* Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all available anti-microbial drugs or intolerance to IV hydration due to pre-existing pulmonary or cardiac impairment
* Subjects with pleural effusion requiring thoracentesis or ascites requiring paracentesis within 14 days prior to admission
* Uncontrolled psychiatric condition
* Any other clinically significant medical or psychiatric disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2020-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Attaphol Pawarode, M.D., Principal Investigator — University of Michgan Cancer Center
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two patients who consented never began treatment.
Groups:
- Dose Level 1 - Maximum Dose Carfilzomib 20 mg/m^2: Participants in all cohorts were administered 20 mg/m^2 of Carfilzomib on days +1 and +2, via intravenous catheter (IV) over 30 minutes.
  Cohort 1: Participants were administered 20 mg/m^2 of Carfilzomib on days +6 and +7.
  Participants in all cohorts were administered tacrolimus at 0.03 mg/kg continuous infusion over 24 hours, starting on day -3 as standard graft-versus-host disease prophylaxis.
- Dose Level 2 - Maximum Dose Carfilzomib 27 mg/m^2: Participants in all cohorts were administered 20 mg/m^2 of Carfilzomib on days +1 and +2, via intravenous catheter (IV) over 30 minutes.
  Cohort 2: Participants were administered 27 mg/m^2 of Carfilzomib on days +6 and +7.
  Participants in all cohorts were administered tacrolimus at 0.03 mg/kg continuous infusion over 24 hours, starting on day -3 as standard graft-versus-host disease prophylaxis.
- Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2: Participants in all cohorts were administered 20 mg/m^2 of Carfilzomib on days +1 and +2, via intravenous catheter (IV) over 30 minutes.
  Cohort 3: Participants were administered 36 mg/m^2 of Carfilzomib on days +6 and +7.
  Participants in all cohorts were administered tacrolimus at 0.03 mg/kg continuous infusion over 24 hours, starting on day -3 as standard graft-versus-host disease prophylaxis.
- Dose Level 4 - Maximum Dose Carfilzomib 45 mg/m^2: "Participants in all cohorts were administered 20 mg/m^2 of Carfilzomib on days +1 and +2, via intravenous catheter (IV) over 30 minutes.
  Cohort 4: Participants were administered 45 mg/m^2 of Carfilzomib on days +6 and +7.
  Participants in all cohorts were administered tacrolimus at 0.03 mg/kg continuous infusion over 24 hours, starting on day -3 as standard graft-versus-host disease prophylaxis.
Period: Phase I: Max Dose 20 mg/m^2 (Day 1-7)
Arm/Group | Dose Level 1 - Maximum Dose Carfilzomib 20 mg/m^2 | Dose Level 2 - Maximum Dose Carfilzomib 27 mg/m^2 | Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2 | Dose Level 4 - Maximum Dose Carfilzomib 45 mg/m^2
Started (Started carfilzomib) | 3 | 0 | 0 | 0
Completed (Completed all 4 doses of Carfilzomib) | 3 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Phase I: Max Dose 27 mg/m^2 (Day 1-7)
Arm/Group | Dose Level 1 - Maximum Dose Carfilzomib 20 mg/m^2 | Dose Level 2 - Maximum Dose Carfilzomib 27 mg/m^2 | Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2 | Dose Level 4 - Maximum Dose Carfilzomib 45 mg/m^2
Started | 0 | 3 | 0 | 0
Completed | 0 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Phase I: Max Dose 36 mg/m^2 (Day 1-7)
Arm/Group | Dose Level 1 - Maximum Dose Carfilzomib 20 mg/m^2 | Dose Level 2 - Maximum Dose Carfilzomib 27 mg/m^2 | Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2 | Dose Level 4 - Maximum Dose Carfilzomib 45 mg/m^2
Started | 0 | 0 | 4 | 0
Completed | 0 | 0 | 3 | 0
Not Completed | 0 | 0 | 1 | 0
Period: Phase I: Max Dose 45 mg/m^2 (Day 1-7)
Arm/Group | Dose Level 1 - Maximum Dose Carfilzomib 20 mg/m^2 | Dose Level 2 - Maximum Dose Carfilzomib 27 mg/m^2 | Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2 | Dose Level 4 - Maximum Dose Carfilzomib 45 mg/m^2
Started | 0 | 0 | 0 | 4
Completed | 0 | 0 | 0 | 2
Not Completed | 0 | 0 | 0 | 2
Period: Phase II: Max Dose 36 mg/m^2 (Day 1-7)
Arm/Group | Dose Level 1 - Maximum Dose Carfilzomib 20 mg/m^2 | Dose Level 2 - Maximum Dose Carfilzomib 27 mg/m^2 | Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2 | Dose Level 4 - Maximum Dose Carfilzomib 45 mg/m^2
Started | 0 | 0 | 37 | 0
Completed | 0 | 0 | 36 | 0
Not Completed | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 1 - Maximum Dose Carfilzomib 20 mg/m^2: Participants were administered 20 mg/m^2 of Carfilzomib on days 1, 2, 6 and 7.
- Dose Level 2 - Maximum Dose Carfilzomib 27 mg/m^2: Participants were administered 20 mg/m^2 on days 1 and 2; 27 mg/m^2 of Carfilzomib on days 6 and 7.
- Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2: Participants were administered 20 mg/m^2 on days 1 and 2; 36 mg/m^2 of Carfilzomib on days 6 and 7.
- Dose Level 4 - Maximum Dose Carfilzomib 45 mg/m^2: Participants were administered 20 mg/m^2 on days 1 and 2; 45 mg/m^2 of Carfilzomib on days 6 and 7.
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 - Maximum Dose Carfilzomib 20 mg/m^2 | Dose Level 2 - Maximum Dose Carfilzomib 27 mg/m^2 | Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2 | Dose Level 4 - Maximum Dose Carfilzomib 45 mg/m^2 | Total
Number analyzed (Participants) | 3 | 3 | 41 | 4 | 51
Age, Continuous [Median (Full Range); unit: years] | 32 [29 to 60] | 55 [51 to 61] | 58 [26 to 69] | 60 [53 to 64] | 58 [26 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 22 | 0 | 24
  Male | 2 | 2 | 19 | 4 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 39 | 4 | 49
  Unknown or Not Reported | 0 | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Maximum Tolerated Dose (MTD) of Carfilzomib
Description: Subjects were enrolled on the first dose level (20 mg/m^2), following a standard 3+3 dose escalation. For any given dose level, if none of the 3 subjects developed a treatment-related dose limiting toxicity (DLT), defined per protocol, dose escalation would follow. If a DLT occurred in any given dose level, the cohort would be expanded to 6. Further dose escalation would be made only if DLTs occurred in <2 out of 6 subjects. If >=2 of 6 develop DLTs, dose de-escalation would be made to the previous level. The highest dose level at which no more than one of six participants experience a DLT defines the MTD.
Time Frame: Up to day 28
Population: Phase 1 study participants
Measure: Number; unit: milligrams per square meter (mg/m^2)
Groups:
- Phase 1 Study Participants: Participants in all cohorts were administered 20 mg/m^2 of Carfilzomib on days +1 and +2, via intravenous catheter (IV) over 30 minutes.
  Dose Level 1, 2, 3, 4: Participants were administered 20, 27, 36, or 45 mg/m^2 of Carfilzomib on days +6 and +7, respectively.
  Participants in all cohorts were administered tacrolimus at 0.03 mg/kg continuous infusion over 24 hours, starting on day -3 as standard graft-versus-host disease prophylaxis.
Arm/Group | Phase 1 Study Participants
Number analyzed (Participants) | 14
milligrams per square meter (mg/m^2) | 36

2. Primary Outcome: Phase II: Kaplan-Meier Estimate of the Percentage of Patients Who Are Alive and Have Not Developed Any "Event"
Description: Kaplan-Meier estimate of the percentage of patients who are alive and have not developed relapse/progression of primary disease or clinical grade III-IV acute graft-versus- host disease (GVHD) or chronic GVHD requiring systemic treatment. Subjects who receive all 4 doses of carfilzomib at the maximum tolerated dose level will be considered evaluable for endpoint analysis.
Time Frame: 1 year
Population: Subjects who have received all 4 doses of carfilzomib at the maximum tolerated dose (MTD) level (dose level 3, 36 mg/m^2): 39 subjects total. Note: three subjects who completed 4 doses of carfilzomib at the MTD during the phase 1 portion of the study were included in phase 2 analysis of the primary outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2 IV: Participants were administered 20 mg/m^2 on days 1 and 2; 36 mg/m^2 of Carfilzomib on days 6 and 7.
Arm/Group | Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2 IV
Number analyzed (Participants) | 39
percentage of participants | 31 [17 to 46]

3. Secondary Outcome: Phase II: Kaplan-Meier Estimate for Progression/Relapse-free Survival Time
Description: Time from day 0 to the date of the first progression/relapse. Subjects who receive all 4 doses of carfilzomib at the maximum tolerated dose level will be considered evaluable for endpoint analysis.
Time Frame: Up to 3 years
Population: Subjects who received all 4 doses of carfilzomib at the maximum tolerated dose (MTD) level (dose level 3, 36 mg/m^2): 39 subjects total. Note: three subjects who completed 4 doses of carfilzomib at the MTD during the phase 1 portion of the study were included in phase 2 analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2
Number analyzed (Participants) | 39
percentage of participants
  1 year since transplant | 72 [59 to 89]
  3 years since transplant | 40 [25 to 62]

4. Secondary Outcome: Phase II: Kaplan-Meier Estimate for Overall Survival Time
Description: The time from day 0 to the day of death from any cause. Subjects who receive all 4 doses of carfilzomib at the maximum tolerated dose level will be considered evaluable for endpoint analysis.
Time Frame: Up to 3 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2
Number analyzed (Participants) | 39
percentage of participants
  1 year since transplant | 72 [59 to 87]
  3 years since transplant | 54 [40 to 72]

5. Secondary Outcome: Number of Regimen Related Toxicities (RRTs)
Description: An RTT is defined as an adverse event (AE) that occurs within +37 days after transplant or 30 days after the last dose of carfilzomib (day +7), and is considered to be a direct consequence and a related event as a result of the combination of conditioning chemotherapy, GVHD prophylaxis regimen and carfilzomib.
Time Frame: Up to 30 days post treatment
Population: Subjects who have received at least one dose of carfilzomib were evaluable for toxicities
Measure: Number; unit: Regimen related toxicities
Groups:
- Dose Level 1 - Maximum Dose Carfilzomib 20 mg/m^2 IV: Participants were administered 20 mg/m^2 of Carfilzomib on days 1, 2, 6 and 7.
- Dose Level 2 - Maximum Dose Carfilzomib 27 mg/m^2 IV: Participants were administered 20 mg/m^2 on days 1 and 2; 27 mg/m^2 of Carfilzomib on days 6 and 7.
- Dose Level 4 - Maximum Dose Carfilzomib 45 mg/m^2 IV: Participants were administered 20 mg/m^2 on days 1 and 2; 45 mg/m^2 of Carfilzomib on days 6 and 7.
Arm/Group | Dose Level 1 - Maximum Dose Carfilzomib 20 mg/m^2 IV | Dose Level 2 - Maximum Dose Carfilzomib 27 mg/m^2 IV | Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2 IV | Dose Level 4 - Maximum Dose Carfilzomib 45 mg/m^2 IV
Number analyzed (Participants) | 3 | 3 | 41 | 4
Regimen related toxicities | 4 | 1 | 15 | 6

6. Secondary Outcome: Phase II: Cumulative Incidence of Acute GVHD
Description: The cumulative incidence of acute Graft Versus Host Disease (aGVHD). Events were assigned a severity grade using the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) v. 4.0; lower values indicate least severe and higher values indicate most severe. Grades 2 - 4 and grades 3 - 4 events are reported. Subjects who receive all 4 doses of carfilzomib at the maximum tolerated dose level will be considered evaluable for endpoint analysis.
Time Frame: At day 180 post-transplant; data collected up to 3 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2
Number analyzed (Participants) | 39
percentage of participants
  Acute GVHD grade 2-4 | 32 [21 to 48]
  Acute GVHD grade 3-4 | 15 [7 to 29]

7. Secondary Outcome: Phase II: Cumulative Incidence of Chronic GVHD
Description: The cumulative incidence of chronic Graft Versus Host Disease (GVHD). Subjects who receive all 4 doses of carfilzomib at the maximum tolerated dose level will be considered evaluable for endpoint analysis.
Time Frame: Up to 3 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2
Number analyzed (Participants) | 39
percentage of participants
  cGVHD overall: Day 180 | 2 [0 to 16]
  cGVHD overall: Day 365 | 15 [7 to 31]
  cGVHD overall: Day 1095 | 15 [7 to 31]
  cGVHD Moderate / Severe: Day 180 | 2 [0 to 16]
  cGVHD Moderate / Severe: Day 365 | 10 [4 to 25]
  cGVHD Moderate / Severe: Day 1095 | 10 [4 to 25]
  cGVHD Requiring Systemic Therapy: Day 180 | 2 [0 to 16]
  cGVHD Requiring Systemic Therapy: Day 365 | 7 [2 to 22]
  cGVHD Requiring Systemic Therapy: Day 1095 | 7 [2 to 22]

8. Secondary Outcome: Phase II: Cumulative Incidence of Non-relapse Mortality
Description: The cumulative incidence of non-relapse mortality. Subjects who receive all 4 doses of carfilzomib at the maximum tolerated dose level will be considered evaluable for endpoint analysis.
Time Frame: Up to 3 years
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2
Number analyzed (Participants) | 39
percentage of participants
  Day 180 | 15 [7 to 29]
  Day 365 | 17 [9 to 31]
  Day 1095 | 23 [14 to 39]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected up to 100 days after the last dose of carfilzomib. All-cause mortality includes all patients followed for up to three years after their first dose of carfilzomib; total duration of data collection was 6 years with an average duration of 1.8 years.
Groups:
- Dose Level 1 - Maximum Dose Carfilzomib 20 mg/m^2 IV: Participants in all cohorts were administered 20 mg/m^2 of Carfilzomib on days +1 and +2, via intravenous catheter (IV) over 30 minutes.
  Cohort 1: Participants were administered 20 mg/m^2 of Carfilzomib on days +6 and +7.
- Dose Level 2 - Maximum Dose Carfilzomib 27 mg/m^2 IV: Participants in all cohorts were administered 20 mg/m^2 of Carfilzomib on days +1 and +2, via intravenous catheter (IV) over 30 minutes.
  Cohort 2: Participants were administered 27 mg/m^2 of Carfilzomib on days +6 and +7.
- Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2 IV: Participants in all cohorts were administered 20 mg/m^2 of Carfilzomib on days +1 and +2, via intravenous catheter (IV) over 30 minutes.
  Cohort 3: Participants were administered 36 mg/m^2 of Carfilzomib on days +6 and +7.
- Dose Level 4 - Maximum Dose Carfilzomib 45 mg/m^2 IV: Participants in all cohorts were administered 20 mg/m^2 of Carfilzomib on days +1 and +2, via intravenous catheter (IV) over 30 minutes.
  Cohort 4: Participants were administered 45 mg/m^2 of Carfilzomib on days +6 and +7.
Arm/Group | Dose Level 1 - Maximum Dose Carfilzomib 20 mg/m^2 IV | Dose Level 2 - Maximum Dose Carfilzomib 27 mg/m^2 IV | Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2 IV | Dose Level 4 - Maximum Dose Carfilzomib 45 mg/m^2 IV
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/3 | 18/41 | 2/4
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 25/41 | 4/4
Other Adverse Events (participants affected / at risk) | 3/3 | 0/3 | 16/41 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 - Maximum Dose Carfilzomib 20 mg/m^2 IV (N=3) | Dose Level 2 - Maximum Dose Carfilzomib 27 mg/m^2 IV (N=3) | Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2 IV (N=41) | Dose Level 4 - Maximum Dose Carfilzomib 45 mg/m^2 IV (N=4)
Anaphylaxis (Immune system disorders) | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 0 | 4 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 1
Chills (General disorders) | 1 | 0 | 0 | 0
Colonic hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Corneal ulcer (Eye disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Encephalitis infection (Infections and infestations) | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Fever (General disorders) | 0 | 0 | 1 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 3 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Immune system disorders - Other (Immune system disorders) | 0 | 0 | 9 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 1 | 4 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 3 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Papulopustular rash (Infections and infestations) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1 | 2 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 - Maximum Dose Carfilzomib 20 mg/m^2 IV (N=3) | Dose Level 2 - Maximum Dose Carfilzomib 27 mg/m^2 IV (N=3) | Dose Level 3 - Maximum Dose Carfilzomib 36 mg/m^2 IV (N=41) | Dose Level 4 - Maximum Dose Carfilzomib 45 mg/m^2 IV (N=4)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 5 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 0 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 4 | 0
Edema limbs (General disorders) | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 4 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Immune system disorders - Other (Immune system disorders) | 0 | 0 | 2 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 3 | 0
Mucositis oral (Gastrointestinal disorders) | 3 | 0 | 5 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 3 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Papulopustular rash (Infections and infestations) | 1 | 0 | 0 | 0
Penile infection (Infections and infestations) | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 3 | 0
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0
White blood cell decreased (Investigations) | 0 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT02145403/Prot_SAP_000.pdf